CLINICAL TRIAL: NCT01161147
Title: Comparative Bioavailability Study of Meloxicam 15 mg Tablets (Dr. Reddy's Laboratories Ltd., Generics) Vs. Mobic® 15 mg Tablets (Boehringer Ingelheim Pharmaceuticals Inc.,Usa) in Healthy Male And/Or Female Volunteers Under Fed Conditions- P1CX04002
Brief Title: Bioequivalence Study of Meloxicam Tablets 15 mg of Dr.Reddy's Laboratories Limited Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Group leader-Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P1CX04002
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2004-08

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meloxicam (Experimental): Meloxicam Tablets 15 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Meloxicam
- Mobic (Active Comparator): Mobic Tablets 15 mg of Boehringer Ingelheim Pharmaceuticals Inc
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam — Meloxicam Tablets 15 mg
  Other Names: Mobic Tablets 15 mg

SUMMARY:
The objective of this study is to determine the relative bioavailability of one 15 mg Meloxicam tablet (Dr. Reddy. Laboratories Ltd.,Generics) versus one 15 mg Mobic (meloxicam) Tablet (Boehringer Ingelheim Pharmaceuticals Inc., USA) under fed conditions.

DETAILED DESCRIPTION:
Twenty eight (twenty six study subjects + two alternate subjects)healthy male and/or female subjects participated in an open label, two-period, two-sequence, two- treatment,single dose, two-way crossover study with at least 14 days washout between doses conducted under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be a healthy male or female volunteer.If the volunteer is female. she must demonstrate β-CG levels consistent with the nongravid state at the medical screening visit and at check-in for Period 1 and agree to remain abstinent or use double-barrier contraception (partner using condom and female volunteer using diaphragm, contraceptive sponge, spermicide, or IUD). If the female is post-menopausal or is surgically sterile, she is exempt from this requirement. (Postmenopausal is defined as no menses for the previous 1 year. If cessation of menses is within 18 months, FSH and/or LH must be documented prestudy as elevated into the postmenopausal range.).
2. The subject must be between the ages of 18 - 55 years old (inclusive).
3. The Subject's body mass index (BMI) must be within 19.0 - 30.0 (Kg/m2).
4. The subject must be a non-smoker and not using any nicotine products.
5. The subject must sign the written consent form (Research Subject Information and Consent Form) prior to study entry.
6. The subject must have clinically acceptable results from the screening procedure including blood pressure, heart rate, ECG, physical exam, medical history, hematology, biochemistry, urinalysis. and infection screen (Hepatitis B Antigen, Hepatitis C Antibody, HIV)

Exclusion Criteria:

1. Subjects with a history of clinically significant gastro-intestinal, dermatological, cardiovascular, renal, hematological, neurological, hepatic, pulmonary, or endocrine disease in the last 12 months.
2. Subjects determined by the Investigator to have any medical condition which may affect the absorption, distribution, metabolism or excretion of the investigational product, or that could jeopardize their health or prejudice the results (e.g. history of surgery of the gastro-intestinal tract, except for appendectomy).
3. Subjects with a known allergy to meloxicam (Mobic) or other nonsteroidal anti-inflammatory drugs (NSAIDS) [e.g. Motrin® (ibuprofen), Celebrex® (celecoxib). Vioxx® (rofecoxib). Naprelan® and Anaprox®, (naproxen sodium), Lodine® (etodolac), Cataflam® (diclofenac potassium). Voltaren® and Arthrotec®(diclofenac sodium), etc.].
4. Females who are pregnant, breastfeeding, or are likely to become pregnant.
5. Subjects with any clinically significant illness within four weeks prior to Period 1 dosing.
6. Subjects with a positive saliva alcohol test at check-in for any period.
7. Subjects with a history of alcohol, drug or substance abuse in the past 12 months.
8. Subjects who have used any prescription medication within 14 days of Period 1 dosing or over-the-counter medication within 14 days of Period 1 dosing.
9. Subjects deemed uncooperative or noncompliant.
10. Subjects who have consumed alcohol within 48 hours prior to Period 1 and Period 2 dosing.
11. Subjects who have consumed xanthine-containing products (including caffeine, theobromines, etc.) within 48 hours prior to Period 1 dosing.
12. Subjects who have consumed food or beverages containing grapefruit (e.g. fresh, Canned, or frozen) within 14 days prior to the administration of the study medication.
13. Subjects who have had an abnormal diet within 30 days prior to Period 1 dosing.
14. Subjects who have participated in an investigational drug study or who have donated more than 100 mL of blood within 30 days prior to Period 1 dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Deepen M Patel, M.D., C.C.F.P., Principal Investigator — Allied Research International Inc.
Locations (1):
- Allied Research International Inc., Mississauga, Ontario, Canada